CLINICAL TRIAL: NCT07312253
Title: The Effect of Web-Based Sexual Education and Counselling Provided to Adolescents on Attitudes Towards Sexual Education and Knowledge Levels
Brief Title: Web-Based Sexual Education and Counseling in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Muhammed Burak Bilgin, PhD Candidate, Nursing, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ADO-WEB-SEXED-01
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Sexual Health Education; Adolescent Health; Sexual Health Knowledge
Keywords: Web-based education; Sexual education; Adolescents; Digital counseling; Nursing intervention
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Adolescents who received structured web-based sexual education and counseling through an online platform.
  Interventions: Behavioral: Web-Based Sexual Education and Counseling
- Control Group (No Intervention): Adolescents who did not receive any intervention and continued with routine education.

INTERVENTIONS:
Behavioral: Web-Based Sexual Education and Counseling — A structured web-based sexual education and counseling program delivered through an online platform, including educational modules and counseling content designed to improve adolescents' sexual health knowledge and attitudes toward sexual education.
  Arms: Intervention Group

SUMMARY:
This study aims to evaluate the effect of a web-based sexual education and counseling program on adolescents' attitudes toward sexual education and their level of sexual health knowledge. The study was conducted as a randomized controlled trial with adolescents enrolled in high school. Participants in the intervention group received structured web-based sexual education and counseling through an online platform, while the control group received no intervention. Data were collected using validated scales before and after the intervention. The findings of this study are expected to contribute to the development of effective digital sexual health education programs for adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 14-18 years.
* Enrolled in high school.
* Provided written informed consent (and parental consent where applicable).
* Access to the internet and a digital device.

Exclusion Criteria:

* Adolescents who did not complete baseline measurements.
* Adolescents who declined participation or withdrew during the study.
* Presence of cognitive or communication problems that prevent understanding the educational content.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Attitude Toward Sexual Education | Baseline and 4 weeks after the intervention
  Attitudes toward sexual education will be assessed using the Attitude Toward Sexual Education Scale, developed by Turhan (2015). The scale is a 5-point Likert-type instrument consisting of 15 items and two subscales: Views on the Benefits of Sexual Education and Views on Sexual Health. Total scores range from 15 to 75, with higher scores indicating more positive attitudes toward sexual education. The scale has demonstrated good internal consistency, with a Cronbach's alpha coefficient of 0.86 for the total scale.

SECONDARY OUTCOMES:
Sexual Health Knowledge Test | Baseline and immediately after the intervention
  The Sexual Health Knowledge Test is a 34-item instrument developed to assess adolescents' level of knowledge regarding sexual health. Each item is answered as "True," "False," or "I do not know." Sixteen items are correct statements and eighteen are incorrect. Correct answers are scored as 1 point, while incorrect and "I do not know" responses are scored as 0. Total scores range from 0 to 34, with higher scores indicating greater sexual health knowledge. The reliability of the test was established using the Kuder-Richardson 20 (KR-20) coefficient (0.71).

CONTACTS AND LOCATIONS:
Locations (1):
- Public High School affiliated with the Provincial Directorate of National Education, Siirt, Turkey, Siirt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No